CLINICAL TRIAL: NCT01540864
Title: A 26 Week Randomized, Double-blind, Placebo-controlled Phase 2 Study to Evaluate the Safety and Efficacy of Various Doses of HPP404 on Weight Loss in Overweight or Obese Subjects
Brief Title: A Safety and Efficacy Study of HPP404 on Weight Loss in Overweight or Obese Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: High Point Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HPP404-201
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-08

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Overweight; Body Mass Index
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- HPP404 35 mg (Experimental)
  Interventions: Drug: HPP404
- HPP404 50 mg (Experimental)
  Interventions: Drug: HPP404
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HPP404 — Administered orally once daily for 26 weeks
  Arms: HPP404 35 mg; HPP404 50 mg
Drug: Placebo — Administered orally once daily for 26 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety and effect of HPP404 versus placebo on body weight in overweight or obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) from 30.0 to 39.9 kg/m2, for subjects with no additional co morbidities;
* BMI from 27 to 39.9 kg/m2, for subjects with co morbidities (i.e. dyslipidemia defined as high LDL (≥ 160 mg/dL) or high total cholesterol (≥ 240 mg/dL), or subjects with hypertension)

Exclusion Criteria:

* Systolic blood pressure > 160 mmHg and/or diastolic pressure > 90 mmHg at the Screening Visit without treatment
* History of use of tobacco or nicotine-containing products 180 days prior to Screening visit
* Subjects with type 2 diabetes or fasting blood glucose concentration ≥ 126 mg/dL
* History of appetite or weight modifying surgeries/procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Percent weight loss | Day 1 to Day 182

SECONDARY OUTCOMES:
Number of subjects attaining a 5% or more weight loss | Day 1 to Day 182
Absolute and percent change in Body Mass Index (BMI) | Day 1 to Day 182

CONTACTS AND LOCATIONS:
Overall Officials: Enrikas Vainorius, M.D., Study Director — High Point Pharmaceuticals, LLC.
Locations (10):
- United States (10):
  - Site 11, Augusta, Georgia
  - Site 3, Valparaiso, Indiana
  - Site 12, Louisville, Kentucky
  - Site 9, Hyannis, Massachusetts
  - Site 10, Saint Paul, Minnesota
  - Site 2, New York, New York
  - Site 1, Charlotte, North Carolina
  - Site 5, High Point, North Carolina
  - Site 7, Norfolk, Virginia
  - Site 6, Richmond, Virginia